CLINICAL TRIAL: NCT05615662
Title: Hybrid Type-1 Effectiveness-implementation Trial for Primary Care Depression Screening and Referral to a Remote Digital Mental Health Clinic
Brief Title: Meru Health Program to Treat Depression in Primary Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of grant funding.
Sponsor: Meru Health, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Curebase Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-MERU-116; R44MH126836 (NIH)
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Depression; Anxiety
Keywords: Mental Health; Digital Mental Health; Depression; Anxiety; Meru Health
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meru Health Program (Experimental): This group of participants will receive the app-based 12-Week Meru Health Program as their study intervention.
  Interventions: Behavioral: Meru Health Program
- Treatment as Usual (Active Comparator): This group of participants will receive "Treatment as Usual" mental health services under the direction and referral of their Primary Care Physician.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Meru Health Program — The Meru Health Program is a 12-week, evidence-based, smartphone-delivered, therapist-supported digital mental health intervention with as-needed psychiatrist oversight. Enrolled participants work through the program with a cohort of peers similarly affected by depression, with whom they can engage in confidential, anonymous, voluntary group chats overseen by a licensed clinical therapist. The MHP incorporates a continuous care model including daily interaction with a dedicated clinician, several evidence-based treatment components such as cognitive behavioral therapy (CBT), behavioral activation therapy, and mindfulness meditation (MM), as well as promising newer types of depression treatments such as HRVB, nutritional psychiatry, and sleep training. Practices are introduced to weekly topics via video lessons that are reinforced via CBT practices, meditations, and biofeedback sessions and therapist messaging.
  Arms: Meru Health Program
Behavioral: Treatment as Usual — Treatment as Usual in this study will include all of the regular standards of care for mental health needs. These standards of care may include, but are not limited to psychotherapy, pharmacotherapy, or complementary therapy.
  Arms: Treatment as Usual

SUMMARY:
Meru Health Inc. seeks to further validate the Meru Health Program (MHP) as a single solution to screening, referral, and treatment in primary care as compared to treatment as usual using a Randomized Controlled Trial (RCT) study design. The goal of this study is to determine the feasibility, effectiveness, and implementability of this digital mental health (DMH) solution.

If proven effective and implementable, more widely integrating the MHP into primary care has the potential to improve the systems of screening, referral, and treatment for depression nationwide. This, in turn, will serve as a solution to improve access to effective care for the millions of Americans currently suffering from depression, ultimately reducing its public health burden.

DETAILED DESCRIPTION:
The goal of this study is to test the MHP as a 'package solution' of screening and treatment in a primary care setting through a 2-step clinical trial process: (1) A smaller proof-of-concept (POC) trial to provide guidance and establish the settings and assessments for (2) A larger confirmatory type 1 hybrid effectiveness Randomized Controlled Trial (RCT) followed by the collection of potential facilitators and barriers to the treatment's wide scale implementation.

The POC study is aimed to develop all of the study materials for the RCT, and test the screening, referral, and study enrollment procedures. 30 participants will be recruited from 1 primary care clinic. The first 15 eligible participants will be referred to TAU, while the second 15 eligible participants will be referred to the MHP. Study assessments will be performed at the baseline (prior to treatment), 6-week, and 12- week (EOT) time points. In addition, at the end of the 12- week study period, we will interview the participants and providers about their experiences with the study to inform the eventual trial. Feedback will be incorporated into improved study methods.

The 300 participant RCT will be used to demonstrate long lasting and significant improvements of the MHP on participants, measured by a set of assessments completed 6 times for each enrolled participant. Study assessments will be performed at the baseline (prior to treatment), 6-, and 12 weeks (EOT) after baseline, as well as 1-, 3-, 6- and 12-month follow-up time points. Using a stepped-wedge randomization study design, 150 participants will be assigned to MHP and 150 to TAU. Participants with a screening PHQ-9 of 10+ will be randomly assigned to MHP or TAU. For TAU participants, primary care providers will not be directed on how to manage the case, while participants in the MHP group will be scheduled into groups of 10-15 individuals who will work through the program together. Participants will receive the Heart Rate Variability Biofeedback (HRV-B) device and be directed to download and follow the MHP app which prompts daily practices and chat communication. Study assessments for both groups will be administered online with response as the primary outcome.

Lastly will be a multistakeholder process evaluation of the delivery of the MHP intervention. Data collected from the 300 RCT participants, as well as administrators and providers from the 8 primary care clinics, will be evaluated for completion rates, engagement metrics, and satisfaction using multiple factors. We will then evaluate the program through surveys and interviews and examine patterns of mental health treatment utilization during the 12-week period, intervention fidelity and competence, attitudes, competencies, and barriers and facilitators of implementation of the MHP.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 score of 10 or more at the time of screening
* Willing to commit to the Meru Health Program if selected
* Proficient in the English language
* At least 18 years of age at the time of enrollment
* Has a valid mailing address
* Owns an Apple or Android smartphone with 1 of the 3 most recent versions of the operating system software.

Exclusion Criteria:

* Active suicide intent with plan to act
* Substance use disorder in the past 3 months
* Ever been diagnosed with bipolar disorder
* Ever been diagnosed with a psychotic disorder
* Currently pregnant
* Less than 3 months postpartum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 scores | Baseline, Week 6, Week 12, 1 Month Follow-up, 3 Month Follow-up, 6 Month Follow-up, 1 Year Follow-up
  This 9-item Questionnaire is to measure levels of depression and is scored from 0-27. Higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder-7 scores | Baseline, Week 6, Week 12, 1 Month Follow-up, 3 Month Follow-up, 6 Month Follow-up, 1 Year Follow-up
  This 7-item Questionnaire is to measure levels of anxiety and is scored from 0-21. Higher scores indicate more severe symptoms.
Change in EUROHIS- Quality of Life-8 scores | Baseline, Week 6, Week 12, 1 Month Follow-up, 3 Month Follow-up, 6 Month Follow-up, 1 Year Follow-up
  This 8-item Quality of Life measurement tool is scored from 5-40. Higher scores indicate a higher satisfaction with life.
Change in PROMIS: Self-Efficacy for Managing Chronic Conditions and Emotions scores | Baseline, Week 6, Week 12, 1 Month Follow-up, 3 Month Follow-up, 6 Month Follow-up, 1 Year Follow-up
  This 4-item Questionnaire is used to measure management of stress and emotions. It is scored from 0-20 with higher scores indicating more severe symptoms.
Change in PROMIS: Sleep Disturbance scores | Baseline, Week 6, Week 12, 1 Month Follow-up, 3 Month Follow-up, 6 Month Follow-up, 1 Year Follow-up
  This 4-item Questionnaire is used to address sleep quality. It is scored from 0-20 with higher scores indicating more severe symptoms.
Change in PROMIS: Sleep-Related Impairment scores | Baseline, Week 6, Week 12, 1 Month Follow-up, 3 Month Follow-up, 6 Month Follow-up, 1 Year Follow-up
  This 4-item Questionnaire is used to address how sleepy a person is during the day and how it affects productivity. It is scored from 0-20 with higher scores indicating more severe symptoms.
Change in Brief Resilience Scale scores | Baseline, Week 6, Week 12, 1 Month Follow-up, 3 Month Follow-up, 6 Month Follow-up, 1 Year Follow-up
  This 6-item Questionnaire is used to measure resilience. It is scored from 1-5 with higher scores indicating greater levels of resilience.
Change in Worker Productivity and Activity Impairment responses | Baseline, Week 6, Week 12, 1 Month Follow-up, 3 Month Follow-up, 6 Month Follow-up, 1 Year Follow-up
  This qualitative questionnaire is used to assess presenteeism, absenteeism, overall worker productivity, and activity impairment. Responses will be analyzed over time to study the employment status, time missed or spent at work, and the impact of health-related issues.
Change in Single Item Burnout responses | Baseline, Week 6, Week 12, 1 Month Follow-up, 3 Month Follow-up, 6 Month Follow-up, 1 Year Follow-up
  This 1-item Questionnaire is used to measure levels of work-related burnout. The responses to this single item will be analyzed over time to study changes in the severity of worker burnout.
System Usability Scale | Week 12
  This 10-item scale that has been validated as a measure of acceptability and satisfaction with digital interventions. It is scored from 0-100, with higher scores indicating higher user satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Peiper, PhD, MPH, Principal Investigator — Meru Health: Director of Research
Locations (1):
- Online Digital Mental Health Clinic, Denver, Colorado, United States